CLINICAL TRIAL: NCT06399172
Title: OncoSil Pancreatic Cancer Post-marketing Clinical Registry Italy
Brief Title: OncoSil Pancreatic Cancer Post-marketing Clinical Registry - Italy
Acronym: OSPRItaly
Status: Not yet recruiting | Type: Observational
Sponsor: OncoSil Medical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: OSPRItaly01
Record Dates: First submitted 2024-04-23; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OncoSil — Intra-tumoural implantation

SUMMARY:
The OSPRItaly Patient Registry has been developed to assess the performance and safety of the OncoSil™ device when used within the approved indication of unresectable, locally advanced pancreatic cancer, in combination with gemcitabine-based chemotherapy, within a real-world observational registry.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are eligible for and undergo OncoSil™ implantation at an eligible treatment facility according to the approved OncoSil™ System Instructions for Use (IFU), as part of their clinical care.
2. Patients who have completed and signed the Patient Informed Consent Form (PICF) for the OSPRItaly Patient Registry.

Exclusion Criteria:

1. Patients participating in an interventional clinical study (company or investigator-sponsored).
2. Use of an investigational agent at the time of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the participating institutions every patient who is intended to undergo implantation of the OncoSil™ device when used within the approved indication of unresectable, locally advanced pancreatic cancer, in combination with gemcitabine-based chemotherapy, in the commercial (sales) setting will be approached by the Principal Investigator (or delegate) to consent to participate in the OSPRItaly Patient Registry.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Followed to death or to 24-months after the date of the last enrolled patient.
  The analysis for safety within the real-world setting will be performed. The safety of OncoSil™ is defined by the Adverse Event profile. All safety summaries will be produced for the Intention-To-Treat (ITT) population. Adverse Device Effects will be coded using Medical Dictionary for Regulatory Activities (MedDRA). All Adverse Device Effects recorded during the Registry will be listed.
  Summary tables will be produced for Treatment Emergent Adverse Device Effects (TEADEs). The number and percentage of patients with device-related Adverse Events by system organ class (SOC) and preferred term will be tabulated. Similar summaries will be produced by severity of event (both mild, moderate or severe, CTCAE grade 1-4) and device relationship.
  In addition, summary tables will be produced for serious TEADEs and TEADEs associated with special interest acute/late radiation effects and or withdrawal.
Tumour response | 1 year
  Target (implanted) tumour response (local and distant)
Device implantation Performance | 1 year
  Safety of the implantation of OncoSil™ within the target tumour will be measured by means of procedure-related Adverse Events. Ease of administration and implantation related data from user questionnaires will be assessed.
Overall Survival | Followed to death or to 24-months after the date of the last enrolled patient
  Overall survival (OS) is defined as the time from enrolment to the date of death from any cause. Patients who are alive or permanently lost to follow-up at the cut-off date for the analysis will be censored at the last date the patient was known to be alive.
Resection Rates | Followed to death or 24 months after the date of the last enrolled patient
  Surgical resection rates and outcome

IPD SHARING:
Plan to Share IPD: No